CLINICAL TRIAL: NCT02986438
Title: Effects of Transcranial Magnetic Stimulation on Functional Connectivity and Response to Treatment of Cocaine Dependent Patients
Brief Title: Treatment With Transcranial Magnetic Stimulation for Cocaine Addiction: Clinical Response and Functional Connectivity.
Acronym: TMS_COC_CONN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Jorge J. González Olvera, Principal Investigator, Instituto Nacional de Psiquiatría Dr. Ramón de la Fuente
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC16036.0
Record Dates: First submitted 2016-12-02; First posted 2016-12-08 (Estimated); Last update posted 2020-07-02 (Actual); Status verified 2020-06

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine; Addiction; rTMS; fMRI
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Double-blind randomized control trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active rTMS frequency at 5 Hz (Active Comparator): The intervention will be Repetitive Transcranial Magnetic Stimulation. Each patient will receive treatment stimulation in the left dorsolateral prefrontal cortex (lDLPFC) with a frequency of 5 Hz, that includes 2 sessions per day for 10 consecutive business days for 2 weeks. Then a target frequency will be determined for the remaining of the study. If this arm's target frequency is chosen, then the participants will receive the maintenance intervention of 2 sessions per week for 12 months. Each session will consist of the application of rTMS at a frequency of 5Hz, to 100% of the motor threshold.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS frequency at 5 Hz (Sham Comparator): The intervention will be Repetitive Transcranial Magnetic Stimulation (Sham). rTMS will be used with a coil that allows simulated stimulation (Coil AP) at a frequency of 5 Hz, with the software necessary for the operator to remain blind to the stimulation condition. This arm will only last for 2 weeks.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (Sham)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — The investigators will use a Magpro R-30 MagVenture quick stimulator, equipped with an 8-reel, 75 mm internal diameter in each spiral.
  Each patient will receive consistent treatment in 2 sessions a day for 10 consecutive business days in the first two weeks, then receive 2 weekly sessions, until the year of treatment is completed. Each session will consist of the application of 30 trains of 10 seconds duration separated by intervals of one minute, at a fixed frequency (5Hz or 10Hz), to 100% of the motor threshold.
  Arms: Active rTMS frequency at 5 Hz
Device: Repetitive Transcranial Magnetic Stimulation (Sham) — The investigators will use a Magpro R-30 MagVenture quick stimulator, equipped with an 8-reel, 75 mm internal diameter in each spiral with a coil that allows simulated stimulation (Coil AP).
  This condition will only last two weeks.
  Arms: Sham rTMS frequency at 5 Hz

SUMMARY:
The purpose of this study is to investigate the short and long term clinical and cognitive effects of repetitive Transcranial Magnetic Stimulation (rTMS) at 5 Hz and/or 10 Hz frequencies on the left dorsolateral prefrontal cortex in cocaine dependent patients and to examine possible changes in brain structure and functional connectivity associated with this intervention.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) has been shown to reduce craving in cocaine addicts in the short term. However, there are no studies on the long term clinical and cognitive effects of sustained rTMS therapy. Moreover, clinical improvement or decline could be related to long term changes in brain structure and function. The purpose of this study is to investigate the short and long term clinical and cognitive effects of repetitive Transcranial Magnetic Stimulation (rTMS) at 5 Hz and/or 10 Hz frequencies on the left dorsolateral prefrontal cortex in cocaine dependent patients and to examine possible changes in brain structure and functional connectivity associated with this intervention. For this purpose the investigators will recruit cocaine dependent patients and stimulate them using rTMS with a acute intervention (twice a day for 2 weeks) and a maintenance intervention (twice a week for 3 months). The investigators will follow the patients to determine clinical outcome. The investigators will also measure clinical, cognitive and brain structural and functional connectivity to asses changes related to the intervention in the short and long term (measurements at: baseline, 2 weeks and 3 months).

Procedure:

The projects consists of: Screening Visit, Part 1 and Part 2.

First, there will be a screening visit, where a clinical interview will be conducted and tests will be applied to select study participants who meet the inclusion and exclusion criteria.

Baseline clinical, cognitive and neuroimaging data will be acquired. The cognitive and neuroimaging data will be exploratory, to be associated with the outcome measures. Part 1 of the study entails the determination of the rTMS target frequency (5 or 10 Hz) for Part 2 (long term stimulation). In Part 1, all participants will be randomly assigned to one of the four treatment legs with rTMS (10Hz, 10Hz-Sham, 5Hz, 5Hz-Sham). Participants will receive 20 sessions of rTMS (intervention or sham), twice per day for 10 consecutive days. Each session lasts approximately 35 minutes.

At 2 weeks, the investigators will evaluate the short term effect of treatment by measuring clinical, cognitive and neuroimaging changes and select which frequency of stimulation is the most effective in terms of clinical improvement, but also in terms of the rate of secondary effects. Our hypothesis is that 5 Hz is as effective as 10 Hz without the high rate of secondary effects (i.e. seizures).

In Part 2 of the study, the sham groups will end and they will be invited to the treatment condition although they data not will be considered for later phases. Here the maintenance phase starts (long term), where rTMS will be performed twice a week for 12 months using the target frequency (5 or 10 Hz). Clinical, cognitive and neuroimaging data will be acquired at 2 weeks and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of eighteen and maximum of fifty years.
* Cocaine users for at least 1 year, currently using at least 3 times a week, with abstinence periods continuing to be less than one month in the last year.
* The reading level of at least 6th grade of primary (equivalent to fifth grade of elementary school).
* The ability to give a valid informed consent.
* Right-handed (in order to control by cerebral laterality in Neuroimaging).
* If the subject is female and of childbearing age, she agrees to use a medically acceptable form of contraception, and to not become pregnant during the duration of the study. A woman is considered to have potential for pregnancy, unless she is postmenopause or surgically sterilized. Female patients of childbearing potential should use either: (1) contraceptive pill or hormone preparation IUD or deposit (ring, injection, implant); And / or (2) a barrier method of contraception, such as the diaphragm, spermicide sponge, or a condom.

Contraceptive measures will be reviewed with the female subjects at each visit prior to the rTMS treatment.

* Self-report of experiencing cocaine craving when exposed to cocaine-associated cues.
* Body mass index less or equal to 30, allowing them to safely enter the Magnetic Resonance.

Exclusion Criteria:

* Personal or first-degree family history of any clinically defined neurological disorder, including organic brain disease, epilepsy, brain events, brain injury, or multiple sclerosis; Or personal history of previous neurosurgery or traumatic brain injury that have produced loss of consciousness.
* Cardiac pacemakers, neural stimulators, implantable defibrillators, implanted medication pumps, intracardiac lines, or acute, unstable heart disease, with intracranial implants (eg, aneurysm clips, leads, stimulators, cochlear implants, or electrodes) or with any other Metallic object inside or near the head that can not be safely removed.
* Screw metal or metallic projectiles into the head or body.
* Current use of any investigational drug or any anti-proconvulsant drug such as tricyclic or neuroleptic antidepressants (which reduce the seizure threshold).
* Increased intracranial pressure (decreasing seizure threshold).
* History of schizophrenia, bipolar disorder, mania or hypomania.
* History of myocardial infarction, angina pectoris, congestive heart failure, cardiomyopathy, cerebrovascular events or transient ischemic attack, or any heart condition currently under medical care.
* Women with reproductive potential who do not use an acceptable form of contraception pregnant or who are lactating.
* Any history of seizures.
* The current dependence (DSM-V criteria) on substances other than cocaine and / or nicotine.
* Claustrophobia making them unable to tolerate lying inside the MRI scanner.
* History of HIV infection or HIV antibody test positive (Due to potential neuroinfection).

These data will be corroborated by a screening visit where the following instruments will be used:

Clinical Interview. Self-applicable demographic questionnaire. Mini International Neuropsychiatric Interview (MINI-Plus). Structured clinical interview for DSM Axis II, self report (SCID-II).

Elimination criteria:

The participation of all participants during the study will be suspended if:

* They express their desire to stop participating.
* They present abnormal radiological findings that require more attention outside the study to ensure the health of the participant.
* Worsening of clinical condition.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Cocaine Craving (CCQ) | Baseline, 2 weeks, 3 months
  The craving will be measured using a craving questionnaire for cocaine validated in Mexican population (Cocaine Craving Questionnaire or CCQ).
Change in Cocaine Craving (VAS) | Baseline, 2 weeks, 3 months
  The craving will be measured using a 100 mm visual analogue scales (VAS).
Change in Cocaine Urine Test | Baseline, 2 weeks, 3 months
  Frequency of cocaine use will be measured using reagent strips from Instant View drug screening (> 300 ng/mL). Results are Positive or Negative.

SECONDARY OUTCOMES:
Changes in Psychopathological Symptoms | Baseline, 2 weeks, 3 months
  Measured by the 90 Symptoms Questionnaire (SCL-90).
Changes in Depression | Baseline, 2 weeks, 3 months
  Measured by Hamilton Depression Rating Scale (HDRS) (21 items).
Changes in Anxiety | Baseline, 2 weeks, 3 months
  Measured by Hamilton Anxiety Rating Scale (HARS).
Changes in Drug Consumption and Related Problems | Baseline, 2 weeks, 3 months
  Measured by the Addiction Severity Index (ASI-lite).
Changes in Sleep Quality: PSQI | Baseline, 2 weeks, 3 months
  Measured by the Pittsburgh Sleep Quality Index (PSQI).
Changes in Impulsivity | Baseline, 2 weeks, 3 months
  Measured by the Barrat Impulsivity Scale-11 (BIS-11).
Lapse rate | Baseline, 2 weeks, 3 months
  Lapse is defined as at least one consumption event not in the same pattern as the baseline consumption. The report of self-consumption of cocaine and urine drug tests, with special attention to the presence of traces of cocaine.
Relapse rate | Baseline, 2 weeks, 3 months
  Relapse is defined as consumption events in the same pattern as the baseline consumption. The report of self-consumption of cocaine and urine drug tests, with special attention to the presence of traces of cocaine.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo A Garza-Villarreal, MD, PHD, Principal Investigator — Universidad Nacional Autonoma de Mexico; Ruth Alcala-Lozano, MD, MSc, Principal Investigator — Instituto Nacional de Psiquiatria "Ramon de la Fuente Muñiz"
Locations (1):
- Instituto Nacional de Psiquiatría "Ramón de la Fuente Muñiz", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
After the main publications by the group are released, all data (clinical, cognitive and neuroimaging) will be uploaded to an online open server such as LONI or OpenfMRI, for example.

REFERENCES:
- [Derived] Garza-Villarreal EA, Alcala-Lozano R, Fernandez-Lozano S, Morelos-Santana E, Davalos A, Villicana V, Alcauter S, Castellanos FX, Gonzalez-Olvera JJ. Clinical and Functional Connectivity Outcomes of 5-Hz Repetitive Transcranial Magnetic Stimulation as an Add-on Treatment in Cocaine Use Disorder: A Double-Blind Randomized Controlled Trial. Biol Psychiatry Cogn Neurosci Neuroimaging. 2021 Jul;6(7):745-757. doi: 10.1016/j.bpsc.2021.01.003. Epub 2021 Jan 26. PMID 33508499